CLINICAL TRIAL: NCT06613165
Title: Exploring the Treatment Duration of PD-1 Neoadjuvant Therapy in Stage II-III dMMR Rectal Cancer: a Prospective，Multicentre, Single-arm Study
Brief Title: Exploring the Treatment Duration of PD-1 Neoadjuvant Therapy in Stage II-III dMMR Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJ dMMR CRC PD-1
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: Immune-related Adverse Event; Neoadjuvant Therapy; dMMR Colorectal Cancer
Keywords: Colorectal Cancer; deficient Mismatch Repair; locally advanced; immune checkpoint
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the optimal number of cycles of PD-1 monotherapy required at minimum, under the premise of ensuring pathological complete response (pCR) among patients with dMMR/MSI-H rectal cancer.

Participants will receive preoperative monotherapy with PD-1 antibodies, with regular reassessments every 2 cycles. Surgical intervention will be performed if clinical complete response (cCR) is achieved.

Researchers will compare the pathological complete response rates, adverse reactions, and three-year event-free survival rates across different treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age: 18 to 80 years old, male or female;
* 2.Patients with histologically or cytologically confirmed dMMR/MSI-H rectal adenocarcinoma, clinical stage II-III;
* 3.No prior systemic therapy, including chemotherapy, radiotherapy, immunotherapy, or targeted therapy;
* 4.ECOG Performance Status (PS) score of 0-1;
* 5.Estimated life expectancy of ≥ 3 months;
* 6.Normal function of major organs, with no severe abnormalities in blood, heart, lung, liver, kidney, bone marrow, or immunodeficiency. Laboratory tests must meet the following criteria: Hemoglobin (Hb) ≥ 90 g/L; White blood cell count (WBC) ≥ 3.0 × 10^9/L; Neutrophil count (NEUT) ≥ 1.5 × 10^9/L; Platelet count (PLT) ≥ 90 × 10^9/L; Liver function (Aspartate Aminotransferase AST or Alanine Aminotransferase ALT) ≤ 2.5 times the upper limit of normal (ULN); Renal function (serum creatinine sCr) ≤ 1.5 times ULN; Total bilirubin (TBIL) ≤ 1.5 times ULN; Urine protein and occult blood < 2+; Fecal occult blood < 2+;
* 7.Subjects must voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up visits;
* 8.The investigator believes that the patient can benefit from the treatment. Physical status score PS ≤ 2;
* 9.Patients and their families must understand and be willing to participate in this study, providing written informed consent.

Exclusion Criteria:

* 1.Patients with a confirmed allergy to the investigational drug and/or its excipients;
* 2.Subjects who have received or are currently receiving additional chemotherapy, radiotherapy, targeted therapy, or immunotherapy;
* 3.Patients with any active autoimmune disease or a history of autoimmune disease;
* 4.Patients with Lynch syndrome;
* 5.Patients with poorly controlled cardiac symptoms or diseases, such as New York Heart Association (NYHA) Class II or higher heart failure, unstable angina pectoris, or myocardial infarction within the past year;
* 6.Pregnant or lactating women;
* 7.Patients with acute infections requiring antibiotic treatment;
* 8.Patients with positive hepatitis B or hepatitis C antibodies;
* 9.Patients with positive HIV antibodies;
* 10.Patients with other diseases that the investigating physician considers may affect prognosis and survival;
* 11.Any other conditions deemed inappropriate for participation in this study by the investigating physician.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage II-III dMMR rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Three-year event-free survival | 2028.09
  Three-year event-free survival (EFS) is a medical metric used in oncology to evaluate the duration over which patients with a particular cancer diagnosis remain free from any cancer-related events, such as disease progression, recurrence, or death from the cancer, within a three-year period following the initiation of treatment.

SECONDARY OUTCOMES:
Pathological complete response，pCR | 2026.09
  Pathological complete response (pCR) is a term used in oncology to describe the absence of any viable tumor cells in the resected tissue specimen following treatment, typically neoadjuvant therapy (such as chemotherapy, radiation therapy, or immunotherapy) prior to surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China